CLINICAL TRIAL: NCT07208929
Title: Investigating Proprioceptive Impairment in Adolescents With Idiopathic Scoliosis (AIS)
Brief Title: Investigating Proprioceptive Impairment in Adolescents With Idiopathic Scoliosis (AIS) (SCOLIO-PROPRIO)
Acronym: SCOLIO-PROPRIO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2025-A00864-45
Record Dates: First submitted 2025-09-17; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Scoliosis Idiopathic Adolescent

STUDY DESIGN:
Intervention Model Description: Propsective, monocentric, comparative study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with Adolescent Idiopathic Scoliosis (Experimental)
  Interventions: Radiation: MRI
- Healthy subjects (No Intervention): External control arm of 30 healthy volounteers from the Human Connectome project from where MRI images will be retrieved.

INTERVENTIONS:
Radiation: MRI — Brain and Spinal Cord MRI
  Arms: Patients with Adolescent Idiopathic Scoliosis

SUMMARY:
The goal of this interventionnal study is to learn if teenagers who have severe scoliosis (a curvature of the spine) have trouble sensing their body's position in space (this sense is called proprioception), which are directly linked to abnormalities in the part of the brain that controls movement and/or caused by the muscles on each side of the spine not being the same size or not developing in the same way.

The main question the investigators aim to answer are :

* Do adolescents with severe scoliosis have problems with their sense of body position (proprioception)?
* If so, are these proprioceptive issues linked to specific problems in the part of the brain that controls movement?
* Are these proprioceptive issues also possibly linked to an uneven muscle structure on either side of the spinal curve?

Researchers will compare the part of the brain that controls movement (ensorimotor brain network) of healthy subjects to that of the participants that will enroll in this study.

Participants will only have to do one more MRI that is not included in the routine of clinical management of scoliosis before surgery.

Data will also be retrieved from clinical practice Participants will answer questionnaires after the day of the surgery

DETAILED DESCRIPTION:
Adolescent Idiopathic Scoliosis (AIS) affects 2 to 4% of the pediatric population. While its exact etiology remains unclear, one leading hypothesis implicates deficits in muscle proprioception, though this remains poorly understood. In addition, structural and functional alterations in brain connectivity have been reported in AIS patients, raising the possibility of a neurobiological underpinning linked to proprioceptive dysfunction.

The primary objective of this study is to determine whether adolescents with severe AIS requiring surgical treatment exhibit structural alterations in the brain's sensorimotor network compared to age-matched control subjects, and whether these alterations are associated with their level of proprioceptive sensitivity. A secondary objective is to assess whether resting-state functional connectivity within the sensorimotor network is also disrupted in AIS patients and whether these functional changes correlate with proprioceptive performance.

The investigators will combine behavioral assessments of static and dynamic proprioception with structural (diffusion MRI) and functional (resting-state fMRI) neuroimaging (using MR scanner at 3T). Static proprioception will be assessed using a joint repositioning test, while dynamic proprioception will be evaluated through vibration-induced movement illusions. This is a prospective, single-center study involving 30 AIS patients and 30 age- and gender-matched healthy controls drawn from open-access neuroimaging databases.

Demonstrating a correlation between brain network alterations and proprioceptive deficits in AIS would provide new evidence in favor of a neuroproprioceptive origin of scoliosis. Such findings could pave the way for the development of targeted proprioceptive rehabilitation strategies in affected adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents diagnosed with Adolescent Idiopathic Scoliosis (AIS) and followed in the pediatric orthopedic surgery department, scheduled to undergo spinal fusion surgery (arthrodesis)
* No history or clinical signs of neurological disorders
* Aged between 10 and 18 years
* Written informed consent obtained from both the adolescent and their legal guardians (parents)
* Control Group only: Participants will be selected from open-access neuroimaging databases, matched to the patient group by age and sex.

Exclusion Criteria:

* Presence of any other clinically significant condition that could be associated with spinal deformity
* Insufficient proficiency in French to understand the informed consent form
* Current treatment with psychotropic medication
* Ongoing pregnancy or breastfeeding
* Subject under legal or judicial supervision
* Contraindications to brain MRI (including: pacemaker; electrically, magnetically, or mechanically activated implants; surgical clips; metallic sutures; staples; etc. - see MRI safety questionnaire annex)
* Subject or their parent(s)/legal guardian(s) refuse to be informed of incidental findings detected during MRI
* Claustrophobia

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between scoliosis and structural brain alteration as assed by dynamic proprioception test and MRI | One day before surgery
  Values of fractional anisotropy (FA) in the corpus callosum and interhemispheric tracts connecting the somatosensory and motor cortices will be compared between the 2 groups of participants
  - The differences found between the two groups (patients versus control) will be correlated to the proprioceptive performances in the patient group as assed by motion illusion amplitude index

SECONDARY OUTCOMES:
Resting state functional connectivity (rs-FC) alteration in AIS assed by MRI | One day before surgery
  We are expecting lower resting-state functional connectivity in patients' sensorimotor network compared to control subjects. We will estimate significant differences in functional connectivity between the 2 groups by comparing connectivity maps
Correlation between Resting-State Functional Connectivity (z-score) as assessed from brain MRI's and Proprioceptive Performance as assessed by measuring the Reproduced Leg Extension Amplitude in degres (°) | Day before surgery
  Identification of the sensorimotor network regions that are most strongly connected in relation to proprioceptive performance by including the illusory range-of-motion index as a co-variate
Correlation between scoliosis gravity as assessed by the cobb angle (°) with previous MRI's and propriovceptive performance as assessed by measuring the Reproduced Leg Extension Amplitude in degres (°) and the quantified gait analysis (°) | One day before surgery
  Dynamic proprioceptive sensitivity - reflected by range-of-motion index - and proprioceptive static sensitivity - reflected by repositioning error - in relation to scoliosis severity estimated on the basis of patients' Cobb angle.
Analysis of scores on body perception as assed by the BESAA | From day one after surgery to 14 day after surgery
  Assessment of body perception by the Body-Esteem Scale for Adolescents and Adults, zero is equivalent to low body perception and 4 is good body perception for each item.
Physical activity as assessed by the Physical Effort Scale (PES) correlated with cobb angle | From day one after surgery to 14 day after surgery
  Physical activity will be assessed by the Physical effort scale will be correlated with the patient's cobb angle retrieved from clinical routine of scoliosis management

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No